CLINICAL TRIAL: NCT01549002
Title: Efficacy of Intranasal Fentanyl at Reducing Pain During Abscess Incision and Drainage (I&D) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Assistant Professor of Clinical Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAI0699
Record Dates: First submitted 2012-02-02; First posted 2012-03-08 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Abscess; Pain
Keywords: Abscess; Pain; Administration intranasal; Infusions intravenous
MeSH Terms: conditions — Abscess; Pain | interventions — Fentanyl; Morphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Fentanyl (Experimental): Patients in this arm will receive intranasal Fentanyl (50 micrograms/mL) as their pre-I&D analgesic. The one time total dose to be used is 2 micrograms / kilogram, to a maximum of 100 micrograms. The medication will be delivered intranasally via an atomizer in 4 equally divided aliquots (2 per nare).
  The abscess I&D will be followed according to protocol using topical and local anesthetic.
  Interventions: Drug: Intranasal Fentanyl
- Intravenous Morphine (Active Comparator): Patients in this arm will receive intravenous morphine as their pre-I&D analgesic. The one time total dose to be used is 0.1 milligrams / kilogram, to a maximum of 8 milligrams. The medication will be delivered via slow IV push.
  The abscess I&D will be followed according to protocol using topical and local anesthetic.
  Interventions: Drug: Intravenous Morphine

INTERVENTIONS:
Drug: Intranasal Fentanyl — Drug: Fentanyl 50 micrograms/mL Dosage: 2 micrograms per kilogram (maximum 100 micrograms) Drug delivery: Intranasal via mucosal atomization device (MAD® Nasal, Wolfe Tory Medical Inc., Salt Lake City, UT) Frequency: one-time dose
  Other Names: Fentanyl
  Arms: Intranasal Fentanyl
Drug: Intravenous Morphine — Drug: Morphine Dosage: 0.1 milligrams/kilogram (maximum 8 milligrams) Drug delivery: Slow IV push Frequency: one-time dose
  Other Names: Morphine
  Arms: Intravenous Morphine

SUMMARY:
Children can develop abscesses (a collection of pus under their skin) that require a physician to cut it open to let the pus drain out. This is a painful procedure. Most medical professionals will use numbing cream and inject numbing medicine into the skin, just like at the dentist, to help reduce the pain. While this helps minimize the pain of cutting the skin, it doesn't help the pain associated with draining out the pus.

There are many strategies and medications available to physicians to help decrease the pain of this procedure. Most of the medications available to treat the pain require the placement of an intravenous (IV) catheter through the patient's skin, which itself is a painful procedure. In the investigators emergency department, many patients with abscesses that need a procedure to drain the pus receive a medicine called morphine through an IV.

Some pain medicines, however, can be sprayed into a patient's nose, and have been shown to be helpful at reducing the pain of a broken bone or a burn. These medicines do not require the placement of an IV.

The purpose of this research study is to determine whether a medicine called fentanyl, when sprayed into the nose of patients aged 4 to 18 years undergoing abscess drainage, is not worse than IV morphine in decreasing the pain of the procedure.

After the risks and benefits of the study are explained to patients and their parents, written informed consent will be obtained. Written informed assent will be obtained for patients older than 8 years of age. Like the flipping of a coin, a computer program will decide randomly which half of the patients will receive fentanyl nose spray and which half will receive morphine by IV.

The patients assigned to receive fentanyl nose spray will not have an IV placed. The patients assigned to receive morphine will have an IV placed. Both groups of patients will have the abscess drainage procedure done the same way. All patients will be videotaped in order to score their pain by a trained observer. This score is the main outcome (measurement) in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 4 years of age up to their 18th birthday
* Patient has a cutaneous abscess for which an I&D is to be performed

Exclusion Criteria:

* Patient's parent doesn't speak English or Spanish
* Patient has developmental delay or neurological impairment
* Patient has altered mental status
* Known hypersensitivity to study drugs (fentanyl, morphine sulfate, lidocaine, LMX4®)
* The presence of significant blood or mucous in the nares despite blowing nose or suctioning
* Severe renal or liver dysfunction, signs of respiratory distress or depression, any respiratory distress, chronic and severe asthma, upper airway obstruction, suspected gastrointestinal obstruction, suspected paralytic ileus
* Narcotic analgesia within 4 hours of ED physician evaluation
* Need for moderate sedation, deep sedation, or general anesthesia
* Need for subspecialty consultation to perform the I&D
* Need for I&D of more than 1 skin abscess
* Cutaneous abscesses located on the genitals, breasts, face, or neck
* Previous enrollment in the study
* Patients with chronic pain syndromes (sickle cell disease, cancer, arthritis, inflammatory bowel disease)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tsze, MD, MPH, Principal Investigator — Columbia University; Peter Dayan, MD, MSc, Study Director — Columbia University; Daniel Fenster, MD, Principal Investigator — Columbia University
Locations (1):
- Alexandra & Steven Cohen Children's Emergency Department of Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Fenster DB, Dayan PS, Babineau J, Aponte-Patel L, Tsze DS. Randomized Trial of Intranasal Fentanyl Versus Intravenous Morphine for Abscess Incision and Drainage. Pediatr Emerg Care. 2018 Sep;34(9):607-612. doi: 10.1097/PEC.0000000000000810. PMID 27387971
- See also: Educational portal for therapeutic intranasal drug delivery — http://www.intranasal.net/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Fentanyl: Patients in this arm will receive intranasal Fentanyl (50 micrograms/mL) as their pre-I&D analgesic. The one time total dose to be used is 2 micrograms / kilogram, to a maximum of 100 micrograms. The medication will be delivered intranasally via an atomizer in 4 equally divided aliquots (2 per nare).
  The abscess I&D will be followed according to protocol using topical and local anesthetic.
  Intranasal Fentanyl: Drug: Fentanyl 50 micrograms/mL Dosage: 2 micrograms per kilogram (maximum 100 micrograms) Drug delivery: Intranasal via mucosal atomization device (MAD® Nasal, Wolfe Tory Medical Inc., Salt Lake City, UT) Frequency: one-time dose
- Intravenous Morphine: Patients in this arm will receive intravenous morphine as their pre-I&D analgesic. The one time total dose to be used is 0.1 milligrams / kilogram, to a maximum of 8 milligrams. The medication will be delivered via slow IV push.
  The abscess I&D will be followed according to protocol using topical and local anesthetic.
  Intravenous Morphine: Drug: Morphine Dosage: 0.1 milligrams/kilogram (maximum 8 milligrams) Drug delivery: Slow IV push Frequency: one-time dose
Period: Overall Study
Arm/Group | Intranasal Fentanyl | Intravenous Morphine
Started | 10 | 10
Completed | 10 | 6
Not Completed | 0 | 4
Not completed — Excessive pain | 0 | 2
Not completed — Moderate sedation required | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Fentanyl | Intravenous Morphine | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15.3 [12.2 to 17.4] | 15.4 [10.2 to 16.4] | 15.4 [11.8 to 16.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 2 | 3 | 5
Observational Scale of Behavioral Distress - revised [Mean (Standard Deviation); unit: units on a scale] — An observational scale of pain and distress during procedures. Scores can range from 0 to 23.5 units for each phase. A higher score indicates a greater degree of pain and distress. The total OSBD-R score is a summation of the OSBD-R score from each phase. For example, if there are six phases, the range of scores for OSBD-R is from 0 to 141. The baseline score would be one of the phases. The baseline phase consisted of 4 15-second intervals. The measured baseline OSBD-R scores was ZERO for all patients.
  units on a scale | 0.06 (0.13) | 0.04 (0.08) | 0.05 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Score on the Observational Scale of Behavioral Distress Revised (OSBD-R)
Description: Our primary outcome is the Observational Scale of Behavioral Distress - Revised (OSBD-R) to assess observed intra-procedural pain. The total OSBD-R score is a summation of the OSBD-R score of each individual phase. The score in each phase can range from 0 to 23.5. There were four phases in our study, so the range of scores for the total OSBD-R was 0 to 94, with a higher score indicating a greater degree of pain and distress. The four phases in the study are (1) before analgesia administration, (2) ten minutes after analgesia administration but before beginning I&D, (3) immediately post I&D procedure (to ascertain the pain perceived during procedure), and (4) ten minutes after procedure completion. The scores documented here are the total OSBD-R scores.
Time Frame: Up to 10 minutes after the procedure completion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Fentanyl | Intravenous Morphine
Number analyzed (Participants) | 10 | 10
units on a scale | 5.48 (4.09) | 18.92 (14.82)

2. Secondary Outcome: Score on the Faces Pain Scale Revised (FPS-R)
Description: The Faces Pain Scale - Revised (FPS-R) is a self-report measure of pain has strong validity and reliability in children 4 - 17 years of age undergoing painful procedures, and will be used to assess patients' self reported pain. A score of 0 means no pain, a score of 10 means very much pain. Therefore, a lower score indicates that a patient is experiencing a lower degree of pain intensity.
  Patients will complete the FPS-R at four times during their medical encounter: (1) before analgesia administration, (2) ten minutes after analgesia administration but before beginning I&D, (3) immediately post I&D procedure (to ascertain the pain perceived during procedure), and (4) ten minutes after procedure completion.
Time Frame: Up to 10 minutes after procedure completion
Population: (1) before analgesia administration, (2) ten minutes after analgesia administration but before beginning I&D, (3) immediately post I&D procedure (to ascertain the pain perceived during procedure), and (4) ten minutes after procedure completion.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intranasal Fentanyl | Intravenous Morphine
Number analyzed (Participants) | 10 | 6
units on a scale
  Before analgesia administration | 6 [3.5 to 6.5] | 4 [1.5 to 6]
  10 min after analgesia, before I&D | 2 [1.5 to 4.5] | 4 [0 to 6]
  Immediately post-I&D | 4 [0 to 8] | 10 [9.5 to 10]
  10 min after procedure completion | 1 [0 to 4] | 5 [2.8 to 6.5]

3. Secondary Outcome: Number of Patients Satisfied With Analgesia Administered
Description: Number of patients satisfied with analgesia administered will be evaluated by determining the number of patients who report a Likert scale response of "somewhat satisfied", "very satisfied", or "extremely satisfied" (i.e. any patient who selects any of these three responses will be considered to have been satisfied with analgesia administered). Patients will be asked 10 minutes after procedure completion. If the patient is 8 years of age and older, both the patient and the parent or guardian will complete a satisfaction survey. If the patients is younger than 8 years, their parent or guardian will complete the satisfaction survey.
Time Frame: 10 minutes after procedure completion
Population: Patient satisfied with analgesia administered
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Fentanyl | Intravenous Morphine
Number analyzed (Participants) | 10 | 10
Participants | 10 | 4

ADVERSE EVENTS:
Description: Standardized cardiopulmonary monitoring and questionnaire.
Arm/Group | Intranasal Fentanyl | Intravenous Morphine
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Fentanyl (N=10) | Intravenous Morphine (N=10)
Oxygen desaturation (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes